CLINICAL TRIAL: NCT03621384
Title: Association of BsmI Polymorphisms in Vitamin D Receptor Gene With Diabetic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Pringgodigdo Nugroho, MD, Head of Dialysis Unit, Dr Cipto Mangunkusumo General Hospital, Indonesia University
Other Study IDs: 756/UN2.F1/ETIK/2014
Record Dates: First submitted 2018-05-22; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Kidney Disease
Keywords: BsmI; Diabetic kidney disease; Polymorphisms; Vitamin D receptor gene
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urea, creatinine, estimated glomerular filtration rate (eGFR), fasting blood glucose (FBG), 2-hours postprandial blood glucose, HbA1c, total cholesterol, triglyceride, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol, BsmI polymorphisms in vitamin D receptor gene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bb Genotype: Subjects with Bb genotype of BsmI polymorphisms in vitamin D receptor gene
- bb Genotype: Subjects with bb genotype of BsmI polymorphisms in vitamin D receptor gene

SUMMARY:
Background: Diabetic kidney disease (DKD), as one of chronic complication of type 2 diabetes mellitus, is common cause of end stage renal disease (ESRD). Vitamin D deficiency is known as one of DKD risk factors. Recent studies on association between vitamin D deficiency and DKD had shown conflicting results. It may be due to vitamin D receptor gene polymorphisms, which is affected by BsmI, Cdx2, ApaI, FokI, and TaqI gene. The investigators conducted cross-sectional study to investigate association between BsmI polymorphisms in vitamin D receptor gene with diabetic kidney disease

Hypothesis: BsmI polymorphisms in vitamin D receptor gene is associated with diabetic kidney disease (DKD)

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD) is a common cause of end stage renal disease (ESRD). Data from Indonesian Renal Registry (2011) revealed that 25% etiology of patients who underwent hemodialysis is DKD. Risk factors that are associated with DKD include blood glucose control, hypertension, dyslipidemia, duration of diabetes mellitus, high body mass index (BMI), age, sex, ethnicity, vitamin D deficiency, high sodium diet, high protein diet, and smoking.

The roles of vitamin D that are related to kidney are inhibition of renin transcription process, angiotensin II, renal inflammation process, and albumin excretion, prevention of podocytes damage, glomerulosclerosis process, and transformation from kidney epithelial cell into mesenchymal cell. Current studies on association between vitamin D deficiency and DKD had shown conflicting results. It may be related to genetic factor which is vitamin D receptor polymorphisms. The vitamin D receptor polymorphism is affected by Cdx2, ApaI, BsmI, FokI, and TaqI gene, where Asian population is mostly affected by ApaI, FokI, and Cdx2.

Several studies had reported the association between BsmI polymorphisms in vitamin D receptor gene and DKD in various population. Zhang, et al (2012) study revealed the association between BsmI polymorphisms in vitamin D receptor gene and DKD in Han Chinese population, while study from Vedralova, et al (2012) in Caucasian race showed opposite result. However, the association between BsmI polymorphism in vitamin D receptor gene and DKD has not been investigated in Indonesian-Malay race.

This is a cross-sectional study that investigate the association between BsmI polymorphisms in vitamin D receptor gene and DKD in Indonesian-Malay race. The investigators collected data about study participants' characteristics, conducted physical examination and laboratory examination, which include BsmI polymorphisms in vitamin D receptor gene.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patient
* Indonesian-Malay race
* Had signed the informed consent

Exclusion Criteria:

* Urinary tract infection
* Pregnant patient
* Fever
* In menstrual period
* Had undergone hemodialysis or peritoneal dialysis
* Had used non steroid antiinflammatory drugs (NSAIDs)
* Postexercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population: type 2 diabetes mellitus patients who live in Indonesia
  Accessible population: type 2 diabetes mellitus patients who visit internal medicine outpatient clinic of dr. Cipto Mangunkusumo Hospital
  Sample: accessible population which meet study criteria
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Association between BsmI Polymorphisms in Vitamin D Receptor Gene and Diabetic Kidney Disease | 1 month
  This study investigated association between BsmI polymorphisms in vitamin D receptor gene with diabetic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Pringgodigdo Nugroho, MD, Principal Investigator — Indonesia University; Suhardjono, Prof., MD, PhD, Principal Investigator — Indonesia University; Aida Lydia, MD, PhD, Principal Investigator — Indonesia University; Kuntjoro Harimurti, MD, PhD, Principal Investigator — Indonesia University; Dekta Filantropi Esa, MD, Principal Investigator — Indonesia University
Locations (1):
- dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Perhimpunan Nefrologi Indonesia. Report of Indonesian Renal Registry. Jakarta; 2011.
- [Result] Ramachandran A, Snehalatha C, Shetty AS, Nanditha A. Trends in prevalence of diabetes in Asian countries. World J Diabetes. 2012 Jun 15;3(6):110-7. doi: 10.4239/wjd.v3.i6.110. PMID 22737281
- [Result] Zhao HL, Thomas GN, Leung W, Tomlinson B, Hsu YH, Chan P. An update on the management of nephropathy in type 2 diabetes. J Chin Med Assoc. 2003 Nov;66(11):627-36. PMID 14768849
- [Result] Tseng CH. Lipid abnormalities associated with urinary albumin excretion rate in Taiwanese type 2 diabetic patients. Kidney Int. 2005 Apr;67(4):1547-53. doi: 10.1111/j.1523-1755.2005.00235.x. PMID 15780110
- [Result] Vedovato M, Lepore G, Coracina A, Dodesini AR, Jori E, Tiengo A, Del Prato S, Trevisan R. Effect of sodium intake on blood pressure and albuminuria in Type 2 diabetic patients: the role of insulin resistance. Diabetologia. 2004 Feb;47(2):300-3. doi: 10.1007/s00125-003-1303-5. Epub 2003 Dec 24. PMID 14704836
- [Result] Dullaart RP, Beusekamp BJ, Meijer S, van Doormaal JJ, Sluiter WJ. Long-term effects of protein-restricted diet on albuminuria and renal function in IDDM patients without clinical nephropathy and hypertension. Diabetes Care. 1993 Feb;16(2):483-92. doi: 10.2337/diacare.16.2.483. PMID 8432221
- [Result] Abbasi MA, Abro A, Sheikh M. Smoking is related to albumin excretion in type 2 diabetes mellitus. Pak J Physiol. 2006;2(2):45-8.
- [Result] Koroshi A, Idrizi A. Renoprotective effects of Vitamin D and renin-angiotensin system. Hippokratia. 2011 Oct;15(4):308-11. PMID 24391410
- [Result] Bid HK, Konwar R, Aggarwal CG, Gautam S, Saxena M, Nayak VL, Banerjee M. Vitamin D receptor (FokI, BsmI and TaqI) gene polymorphisms and type 2 diabetes mellitus: a North Indian study. Indian J Med Sci. 2009 May;63(5):187-94. PMID 19584489
- [Result] Zhang H, Wang J, Yi B, Zhao Y, Liu Y, Zhang K, Cai X, Sun J, Huang L, Liao Q. BsmI polymorphisms in vitamin D receptor gene are associated with diabetic nephropathy in type 2 diabetes in the Han Chinese population. Gene. 2012 Mar 10;495(2):183-8. doi: 10.1016/j.gene.2011.12.049. Epub 2012 Jan 5. PMID 22245613
- [Result] Vedralova M, Kotrbova-Kozak A, Zeleznikova V, Zoubkova H, Rychlik I, Cerna M. Polymorphisms in the vitamin D receptor gene and parathyroid hormone gene in the development and progression of diabetes mellitus and its chronic complications, diabetic nephropathy and non-diabetic renal disease. Kidney Blood Press Res. 2012;36(1):1-9. doi: 10.1159/000339021. Epub 2012 Jun 18. PMID 22777106
- [Result] Dewi K. Penurunan fungsi ginjal pada pasien DM tipe 2 di Poliklinik Endokrin Metabolik RSUPN Cipto Mangunkusumo. University of Indonesia; 2007.
- [Result] Indra T. Asosiasi antara status vitamin D (25(OH)D) dengan albuminuria pada pasien diabetes melitus tipe 2. University of Indonesia; 2013.
- [Result] Giunti S, Barit D, Cooper ME. Mechanisms of diabetic nephropathy: role of hypertension. Hypertension. 2006 Oct;48(4):519-26. doi: 10.1161/01.HYP.0000240331.32352.0c. Epub 2006 Sep 4. No abstract available. PMID 16952978
- [Result] Bayliss G, Weinrauch LA, D'Elia JA. Pathophysiology of obesity-related renal dysfunction contributes to diabetic nephropathy. Curr Diab Rep. 2012 Aug;12(4):440-6. doi: 10.1007/s11892-012-0288-1. PMID 22638939
- [Result] Abbate M, Zoja C, Remuzzi G. How does proteinuria cause progressive renal damage? J Am Soc Nephrol. 2006 Nov;17(11):2974-84. doi: 10.1681/ASN.2006040377. Epub 2006 Oct 11. PMID 17035611
- [Result] Nosratabadi R, Arababadi MK, Salehabad VA, Shamsizadeh A, Mahmoodi M, Sayadi AR, Kennedy D. Polymorphisms within exon 9 but not intron 8 of the vitamin D receptor are associated with the nephropathic complication of type-2 diabetes. Int J Immunogenet. 2010 Dec;37(6):493-7. doi: 10.1111/j.1744-313X.2010.00953.x. Epub 2010 Aug 19. PMID 20727043
- [Result] Inassi J, Vijayalakshmy R. Role of duration of diabetes in the development of nephropathy in type 2 diabetic patients. Natl J Med Res. 2013;3(1):8-11.